CLINICAL TRIAL: NCT05070169
Title: Early Surgical Fixation of Low-Velocity Hip Fractures in Patients With Direct Oral Anticoagulation
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Valerie Weihs, Principal Investigator, Medical University of Vienna
Other Study IDs: 1636/2021
Record Dates: First submitted 2021-09-22; First posted 2021-10-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Surgical Fixation: Prospective cohort of patients with intertrochanteric fractures with DOAC (direct oral anticoagulation) therapy undergoing early surgical fixation (within 24 hours).
  Interventions: Procedure: Early Surgical Fixation vs. Delayed Surgical Fixation
- Delayed Surgical Fixation: Retrospective control group of patients with intertrochanteric fractures with DOAC medication who underwent delayed surgical fixation (≥48 hours) from January 2014 to December 2018.

INTERVENTIONS:
Procedure: Early Surgical Fixation vs. Delayed Surgical Fixation — Evaluation of the reduction of the peri-operative blood loss in patients undergoing early surgical fixation (within 24 hours) of an intertrochanteric fracture under DOAC therapy compared to a retrospectively enrolled group of patients who underwent delayed surgical fixation (≥48 hours) of an intertrochanteric fracture under DOAC therapy.
  Groups: Early Surgical Fixation

SUMMARY:
Prospective cohort study on patients with intertrochanteric fractures under direct oral anticoagulation (DOAC) therapy undergoing early surgical fixation (within 24 hours). The primary aim of this study is to evaluate the reduction of the peri operative blood loss. The secondary aim is to assess the influence of early surgical fixation of intertrochanteric fractures in patients with DOAC therapy on the 30-day and 1-year mortality. Moreover, the prospective cohort group of patients will be compared with a retrospectively analyzed age-, gender- and fracture-type-matched control group of patients who underwent delayed surgical fixation from January 2014 to December 2018 (≥ 48 hours).

ELIGIBILITY:
Inclusion Criteria:

Prospective cohort study:

Patients with intertrochanteric fractures that need a surgical fixation and under treatment with a DOAC medication

Control group:

Patients with intertrochanteric fractures under DOAC medication with a delayed surgical fixation from January 2014 to December 2018 (≥ 48 hours after the trauma)

Exclusion Criteria:

Prospective cohort group:

* patients with multiple fractures
* acute heart failure, kidney and lung failure and
* other concomitant diseases which prevent prompt fixation

Retrospective cohort group:

Patients with delayed surgical fixation due to other causes than DOAC medication (e.g. multimorbidity, acute myocardial infarction, acute heart, lung or kidney failure)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 140 patients with intertrochanteric fractures with DOAC therapy undergoing surgical fixation: 70 patients will be included prospectively starting with October 2021, 70 patients with a delayed surgical fixation will be included retrospectively within the time frame January 2014- December 2018.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the perioperative blood loss | 3 days
  The main objective of this study is the evaluation of the perioperative blood loss in patients with intertrochanteric fractures with DOAC medication treated in a level I trauma center undergoing early surgical fixation (within 24 hours after the trauma). After routine surgical fixation of the fracture, patients will receive blood draws at day 3 according to standardized routinely performed clinical procedures. The perioperative blood loss will be calculated using the "haemoglobin balance method".
Evaluation of the perioperative need for transfusions | 3 days
  The rate of transfusion will be expressed as the percentage of patients who need at least one unit of red blood cells (RBCs) and the total number of transfused RBC units will be recorded. Only perioperative transfusion up to the third post-operative day will be considered.

SECONDARY OUTCOMES:
Coagulation parameters | 3 days
  Coagulation parameters such as plasma DOAC concentrations and Clot Pro analyzes will be measured in accordance with routine clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Traumatology, Vienna, Austria